CLINICAL TRIAL: NCT02568787
Title: The Effect of an Enhanced Rice Bran Nutritional Supplement on Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: The Effect of an RBAC Supplement (BRM4) on NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Daiwa Health Development (Other)
Responsible Party: Principal Investigator, John E. Lewis, Principal Investigator, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20150512
Record Dates: First submitted 2015-10-01; First posted 2015-10-06 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; cytokines; interleukin (IL); interferon (IFN); liver function test (LFTS); nutrition; bran arabinoxylan compound (RBAC); tumor necrosis factor -- type I receptor (TNF-RI); TNF-RII (tumor necrosis factor -- type II receptor (TNF-RII)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rice bran arabinoxylan compound (RBAC) (Experimental): Take 2 tablets 1 time (1 gram) per day for the 3-month intervention period.
  Interventions: Dietary Supplement: rice bran arabinoxylan compound (RBAC)
- Placebo (Placebo Comparator): Take 2 tablets 1 time (1 gram) per day for the 3-month intervention period.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: rice bran arabinoxylan compound (RBAC) — Take 2 tablets 1 time (1 gram) per day for the 3-month intervention period.
  Arms: Rice bran arabinoxylan compound (RBAC)
Dietary Supplement: Placebo — Take 2 tablets 1 time (1 gram) per day for the 3-month intervention period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of Rice Bran Arabinoxylan Compound (RBAC) on outcome variables in persons with non-alcoholic fatty liver disease (NAFLD). This nutritional supplement is made from a water soluble extract of rice bran that has been partially hydrolyzed by the action of a natural enzyme complex extracted from Shiitake mushroom.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of Rice Bran Arabinoxylan Compound (RBAC) on outcome variables in persons with non-alcoholic fatty liver disease (NAFLD). This nutritional supplement is made from a water soluble extract of rice bran that has been partially hydrolyzed by the action of a natural enzyme complex extracted from Shiitake mushroom. Given that these micronutrients may be important for regulating the immune system, investigators will investigate the impact of RBAC on the following variables among 20 adults (18+ years of age and over) diagnosed with NAFLD:

1. albumin
2. 4-hydroxynonenal
3. lipids
4. liver enzymes (alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP)
5. malondialdehyde
6. γ-glutamyltransferase
7. cytokines (TNF-α, LT-α, IL-1α, IL-1β, IL-6, TNF-RI, TNF-RII, IFN-γ, IL-12, IL-2, IL-15, IL-8, IL-4, IL-5, IL-17, IL-23, IL-10, IL-13, and IL-18)
8. lymphocytes
9. platelets

Specifically, subjects will participate in a 3-month, two-group, randomized intervention, where one group (n=10) will take 1 gram/day RBAC and the other group (n=10) will take a placebo to compare differences in outcomes between the two groups. The results of the study are intended to address the multi-faceted physiological problems of NAFLD patients by testing the efficacy of a nutritional supplement intervention on multiple outcomes in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Confirmed NAFLD diagnosis
3. On a stable medication regimen during the intervention
4. Planning to maintain current medication during the course of the intervention
5. Willing to have blood drawn
6. Previous nutritional supplement usage of similar polysaccharide formula permitted, but current use must be stopped 2 weeks before and during trial
7. Interested in participating in a dietary supplement study
8. Willing to follow recommendations for participating in the study
9. Willing to not consume food, alcohol, caffeine, or stimulants (amphetamines) 12 hours before each assessment
10. Able to provide informed consent

Exclusion Criteria:

1. Currently enrolled in another research trial for similar investigative nutritional therapies
2. Known allergy to rice, rice bran, mushrooms, or related food products
3. Any gastrointestinal disorders that could lead to uncertain absorption of the study supplement
4. Taking any lipid-lowering agent for the prior 3 months before study enrollment
5. Currently taking immunomodulatory medication, i.e., interferon
6. Currently taking chemotherapeutic agents
7. Severe anemia or other medical condition that will not permit a safe blood draw
8. A bleeding disorder
9. A terminal illness
10. Women who are pregnant or are attempting conception, especially in the presence of a history of recurrent spontaneous abortion
11. Currently undergoing internal defibrillation, like with an implantable heart device
12. Erratic, accelerated, or mechanically controlled irregular heart rhythms
13. Atrial fibrillation/flutter
14. Atrioventricular block
15. Recently had dyes introduced into the bloodstream, such as methylene blue, indocyanine green, indigo carmine, and fluorescein
16. Any implanted electronic device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06-10 (Actual); Study Completion 2017-06-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in liver function test | Baseline, 45 days and 90 days
  Liver function tests as defined by serum ALT, AST and ALP
Change from baseline in metabolic markers | Baseline,45 days and 90 days
  Metabolic markers as defined by lipid profile
Change from baseline in immunological markers | Baseline,45 days and, 3 months
  Immunological markers as defined by TNF-α, LT-α, IL-1α, IL-1β, IL-6, TNF RI, IFN-γ, IL-12, IL-2, IL-15, IL-8, TNF RII, IL-4, IL-5, IL-17, IL-23, IL-10, IL-13, and IL-18.

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure | Baseline,45 days and 3 months
  Systolic blood pressure will be measured to the nearest even digit by use of the Microlife Deluxe upper arm blood pressure monitor. Three readings will be made with the subjects seated after they have rested for five minutes. The average of the three readings will be used in the analysis.
Change from baseline in Diastolic blood pressure | 45 days and 90 days
  Diastolic blood pressure will be measured to the nearest even digit by use of the Microlife Deluxe upper arm blood pressure monitor. Three readings will be made with the subjects seated after they have rested for five minutes. The average of the three readings will be used in the analysis.
Pulse | Baseline,45 days and 3 months
  Pulse will be measured to the nearest even digit by use of the Microlife Deluxe upper arm blood pressure monitor. Three readings will be made with the subjects seated after they have rested for five minutes. The average of the three readings will be used in the analysis.
Change from Baseline in Quality of Life | Baseline,45 days and 3 months
  The SF-36v2™ Health Survey (15) provides psychometrically-based physical and mental health summary measures and a preference-based health utility index. It is a generic measure that does not target a specific age, disease, or treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: John E Lewis, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Soffer Clinical Research Center, Department of Psychiatry & Behavioral Sciences, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parnell JA, Raman M, Rioux KP, Reimer RA. The potential role of prebiotic fibre for treatment and management of non-alcoholic fatty liver disease and associated obesity and insulin resistance. Liver Int. 2012 May;32(5):701-11. doi: 10.1111/j.1478-3231.2011.02730.x. Epub 2011 Dec 30. PMID 22221818
- [Background] Byrne CD, Olufadi R, Bruce KD, Cagampang FR, Ahmed MH. Metabolic disturbances in non-alcoholic fatty liver disease. Clin Sci (Lond). 2009 Apr;116(7):539-64. doi: 10.1042/CS20080253. PMID 19243311
- [Background] Browning JD, Szczepaniak LS, Dobbins R, Nuremberg P, Horton JD, Cohen JC, Grundy SM, Hobbs HH. Prevalence of hepatic steatosis in an urban population in the United States: impact of ethnicity. Hepatology. 2004 Dec;40(6):1387-95. doi: 10.1002/hep.20466. PMID 15565570
- [Background] Preiss D, Sattar N. Non-alcoholic fatty liver disease: an overview of prevalence, diagnosis, pathogenesis and treatment considerations. Clin Sci (Lond). 2008 Sep;115(5):141-50. doi: 10.1042/CS20070402. PMID 18662168
- [Background] Neuschwander-Tetri BA, Caldwell SH. Nonalcoholic steatohepatitis: summary of an AASLD Single Topic Conference. Hepatology. 2003 May;37(5):1202-19. doi: 10.1053/jhep.2003.50193. PMID 12717402
- [Background] Dowman JK, Armstrong MJ, Tomlinson JW, Newsome PN. Current therapeutic strategies in non-alcoholic fatty liver disease. Diabetes Obes Metab. 2011 Aug;13(8):692-702. doi: 10.1111/j.1463-1326.2011.01403.x. PMID 21449949
- [Background] Patel AA, Torres DM, Harrison SA. Effect of weight loss on nonalcoholic fatty liver disease. J Clin Gastroenterol. 2009 Nov-Dec;43(10):970-4. doi: 10.1097/MCG.0b013e3181b57475. PMID 19727004
- [Background] Musso G, Gambino R, Cassader M, Pagano G. A meta-analysis of randomized trials for the treatment of nonalcoholic fatty liver disease. Hepatology. 2010 Jul;52(1):79-104. doi: 10.1002/hep.23623. PMID 20578268
- [Background] Zheng S, Sanada H, Dohi H, Hirai S, Egashira Y. Suppressive effect of modified arabinoxylan from rice bran (MGN-3) on D-galactosamine-induced IL-18 expression and hepatitis in rats. Biosci Biotechnol Biochem. 2012;76(5):942-6. doi: 10.1271/bbb.110968. Epub 2012 May 7. PMID 22738964
- [Background] Zheng S, Sugita S, Hirai S, Egashira Y. Protective effect of low molecular fraction of MGN-3, a modified arabinoxylan from rice bran, on acute liver injury by inhibition of NF-kappaB and JNK/MAPK expression. Int Immunopharmacol. 2012 Dec;14(4):764-9. doi: 10.1016/j.intimp.2012.10.012. Epub 2012 Oct 29. PMID 23116638
- [Background] Ghoneum M. Enhancement of human natural killer cell activity by modified Arabinoxylan from rice bran (MGN-3). Int J Immunotherapy 1998;14(2):89-99.
- [Background] Ghoneum M, Matsuura M. Augmentation of macrophage phagocytosis by modified arabinoxylan rice bran (MGN-3/biobran). Int J Immunopathol Pharmacol. 2004 Sep-Dec;17(3):283-92. doi: 10.1177/039463200401700308. PMID 15461862
- [Background] Tazawa K, Namikawa H, Oida N, Masada M, Maeda H. Scavenging activity of modified arabinoxylane from rice bran (biobran/mgn-3) with natural killer cell activity on free radicals. Biotherapy 2000;14:493-5.
- [Background] Ali K, Melillo A, Leonard S, Asthana D, Woolger J, Wolfson A, et al. An open-label, randomized clinical trial to assess the immunomodulatory activity of a novel oligosaccharide compound in healthy adults. Functional Foods in Health and Disease 2012;2(7):265-79.
- [Background] Ware J, Kosinski M, Dewey J. How to score version two of the SF-36 health survey. Lincoln, RI: QualityMetric, Incorporated; 2000. ISBN 1891810057